CLINICAL TRIAL: NCT01748123
Title: Creating an Active Collaborative Network of Comparative Effectiveness Researchers: A Randomized Study of Initial Diuretic Therapy for Hypertension.
Brief Title: EBMtrialcentral- Comparing Initial Diuretic Therapies Using a Collaborative Network
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCORI-EGID 4231; 00041242 (Other: Johns Hopkins University)
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Hypertension
Keywords: Pragmatic; Comparative Effectiveness
MeSH Terms: conditions — Hypertension | interventions — Chlorthalidone; atenolol, chlortalidone drug combinations; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorthalidone (Active Comparator): 25mg daily orally for 8 weeks
  Interventions: Drug: Chlorthalidone
- Hydrochlorothiazide (Active Comparator): 50mg daily orally for 8 weeks
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Chlorthalidone — Initial dose of 12.5mg daily Chlorthalidone (force titrated to 25mg at 4 weeks)
  Other Names: Hygroton, Tenoretic
  Arms: Chlorthalidone
Drug: Hydrochlorothiazide — Initial dose 25mg daily HCTZ (force titrated to 50mg at 4 weeks)
  Other Names: Apo-hydro, Aquazide h, Dichlotride, Oretic
  Arms: Hydrochlorothiazide

SUMMARY:
* Clinical equipoise exists with respect to the important question, "What is the best initial diuretic for the treatment of Hypertension"? A pragmatic comparative effectiveness research (CER) study comparing Chlorthalidone to Hydrochlorthiazide (HCTZ) could help inform decision making for this common problem.
* The investigators aim to harness both the power of bioinformatics (using web-based data-capture and electronic health records) and of online media (through collaboration) in order to facilitate such a CER in "usual-care" settings. This process may also provide a foundation for testing a wealth of important clinical questions which commonly arise in the delivery of contemporary healthcare and would otherwise be left unanswered.
* To this end the investigators are developing a website, EBMtrialcentral, where eligible physicians can go online and join their collaborative network. Physicians can then enroll eligible patients in this study. These will include under-served urban patients. Clinical information will be entered online (using a secure database housed at Johns Hopkins), patient consent will be obtained electronically and treatment recommendations will be randomly allocated to either 25mg daily of oral HCTZ or 12.5mg daily of oral Chlorthalidone. The investigators aim to increase to 50mg HCTZ and 25mg Chlorthalidone over 8 weeks and compare their effects on BP measured with a 24 hour monitor.
* The investigators' primary hypothesis is that non-blinded, random, parallel allocation of 12.5mg daily Chlorthalidone (titrated to 25mg at 4 weeks) will demonstrate a clinically meaningful ≥5mmHg improvement in BP control (as measured by change in BP from baseline using 24hr ABPM) compared to 25mg daily HCTZ (titrated to 50mg at 4 weeks) in newly hypertensive patients followed in a usual-care clinic setting over 8 weeks. They will also analyze differences in side-effects or safety (serum electrolytes) between these two medications.

DETAILED DESCRIPTION:
- BACKGROUND:

The application of many traditional randomized controlled trial(RCT) findings to real-world practice is in question. To this end, comparative effectiveness research(CER) has evolved. However, there remains ample evidence that U.S. trials are becoming increasingly cumbersome and expensive. Moreover, 90 percent fail to meet enrollment goals.

In contrast, there have been significant recent technological advances in both bioinformatics and social media. However, thus-far, the combined potential of both has yet to be achieved in the field of medicine. The stage is now set for an amalgamation of these three disciplines; CER, bioinformatics and social media. EBMtrialcentral is a non-profit website developed at Johns Hopkins University with the idea of using an online social network to actually perform CER trials. By harnessing the power of social media, EBMtrialcentral could open up a world of opportunity for conducting clinical research and bring randomization into "usual care".

* OBJECTIVES:

  1. To determine if a social network website can be created, among a group of academic physicians, with the pre-specified objective of using this website to conduct a CER trial.
  2. To perform a pilot-study though the website. This study will randomly allocate initial anti-hypertensive treatment strategies, using guideline recommended diuretic agents.
* METHODS:

  1. Website development-A test website, EBMtrialcentral.org, has been initiated. By visiting the website, eligible physicians will be able to join the collaborative network. Once a member physician identifies an eligible patient who agrees to participate, consent forms will be generated online for formal enrollment. A therapeutic strategy will be randomly allocated via the website. The investigators' platform would require parsimonious imputation of secured patient data. Follow-up will be pragmatic and guideline-directed. Data will initially be managed in a protected online database run by "project REDCap". Patients and patient advocate stakeholders will be invited to help with IRB and website development.
  2. Pilot study-Despite stronger evidence for chlorthalidone, most hypertensive patients prescribed diuretics currently receive HCTZ. However, the two have not been randomly compared in an adequately powered study. The investigators will require 80 newly hypertensive urban subjects to detect a greater than 5mmHg mean automated BP difference between the two groups over 2 monthly follow-up visits (8 weeks total, with a standardized effect size of 0.7 based on prior data). The investigators will include ethnic and under-served subjects. Exclusion criteria will include compelling indications for alternative anti-hypertensives. Non-blinded random allocation will be generated online.

ELIGIBILITY:
Inclusion Criteria:

* Men and women are eligible if they have hypertension, are not receiving antihypertensive medications, and have average office BP values within the last 6 months ≥140/90 mmHg.

Exclusion Criteria:

* Patients with hypertensive urgency will be excluded (BP ≥180/120 mmHg). We also plan to exclude those with "compelling indications" for an Angiotensin Converting Enzyme (ACE) inhibitor or Beta-blocker therapy (per JNC 7). These include those with; a history of diabetes (prior HbA1c ≥6.5%, fasting glucose ≥126mg/dl, a history of insulin or oral hypoglycemic use, or microalbuminuria), myocardial infarction within the last 3 years, and a known LVEF <50%. Other safety exclusions will be; a history of chronic kidney disease (or a serum creatinine ≥1.8 mg/dL), known allergy to study medications, inability to provide consent, a history of significant non-compliance or missed appointments, a history of poorly-controlled gout and a history of falls or autonomic dysfunction and subjects aged <21years or ≥90yrs.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Mean systolic 24 Hour Ambulatory Blood Pressure | 8 weeks

SECONDARY OUTCOMES:
Subjective Medication Side Effects | 4 and 8 weeks

OTHER OUTCOMES:
Serum Potassium | 4 and 8 weeks
  Potassium
Serum Magnesium | 4 and 8 weeks
  Magnesium
Office Systolic BP assessment | 4 and 8 weeks
  Sphygmomanometer

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Schulman, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States